CLINICAL TRIAL: NCT02432482
Title: A Mobile Intervention to Promote Cessation in HIV-infected Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: George Washington University (Other); University of Michigan (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-3094; 1R34DA037042-01 (NIH)
Record Dates: First submitted 2014-10-23; First posted 2015-05-04 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Tobacco Use; HIV-1-infection
Keywords: Tobacco; Cigarette; HIV; Treatment; Mobile; Smartphone
MeSH Terms: conditions — Tobacco Use | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard care (Active Comparator): Brief advice to quit (less than 5 minutes) Self-help brochure Offer of nicotine patches
  Interventions: Behavioral: Standard care
- mobile Positively Smoke Free (mPSF) (Experimental): mPSF: a targeted, intensive behavioral cessation intervention for PLWH smokers
  * offer of nicotine patches
  Interventions: Behavioral: mobile Positively Smoke Free (mPSF)

INTERVENTIONS:
Behavioral: mobile Positively Smoke Free (mPSF) — mPSF is a targeted, intensive behavioral cessation intervention designed for HIV-infected smokers. It is guided by the Social Cognitive Theory model. It includes 8 weekly sessions of audio/video messages to users, daily text messages, and a variety of other smartphone capabilities, e.g. play-a-tune, play-a-game, phone-a-friend, call the quitline.
  Other Names: mPSF
  Arms: mobile Positively Smoke Free (mPSF)
Behavioral: Standard care — Brief advice to quit (<5 minutes) Self-help brochure Offer of nicotine patches
  Other Names: SC
  Arms: Standard care

SUMMARY:
The purpose of this study is to adapt an existing web-based tobacco treatment program for HIV-infected smokers into a mobile intervention delivered via smartphone. After the adaptation is completed, the investigators will test the program's efficacy at promoting abstinence in a randomized controlled trial.

DETAILED DESCRIPTION:
There are nearly one million persons living with confirmed HIV infection (PLWH) in the US, 60% of them smoke cigarettes, and 75% of them are interested in quitting. Almost none are currently accessing smoking cessation interventions designed to meet their specific needs and concerns.

Cigarette smoking is a leading contributor to mortality among PLWH in the HAART era, and it is the direct cause of 30% of non-AIDS defining malignancies. It is driving the alarming rise in cardiac events and lung cancers in this highly vulnerable population. The lack of access to proven, effective, culturally appropriate tobacco cessation services represents a health disparity of the first order. The psychosocial profile of the PLWH-smoker community, characterized by high rates of psychiatric comorbidity, drug and alcohol use, and low levels of social support, suggests that achieving high cessation rates will be a great challenge.

Positively Smoke Free is an intensive, multisession, cessation intervention specifically developed for PLWH smokers. It is currently available as a live, group therapy program and also as a web-based version designed for notebook or desktop computers. In its current form, the web-version is not adoptable to the smartphone platform. Pilot data from randomized, controlled, trials of both formats show promise.

The number of individuals in the US who own smartphones and who use them to access health information on the internet is steadily growing. This growth is most pronounced in the ethnic minority groups that make up the majority of the PLWH community in the US. Behavioral interventions delivered via smartphones offer the advantage of expansive reach, low cost, and immediacy of access to users. A burgeoning body of literature suggests that this may be an especially effective tool for tobacco treatment. mHealth tobacco treatment interventions for PLWH smokers have not yet been explored.

This proposal aims (1) to adapt Positively Smoke Free to the mobile format for smartphones (2) to test the feasibility (i.e. recruitment, adherence, retention, satisfaction, and cost) of mobile Positively Smoke Free (mPSF) in a cohort of 50 PLWH smokers, (3) to complete a pilot randomized controlled trial comparing biochemically confirmed 3-month abstinence rates in subjects (N=50) assigned to the mPSF condition versus those (N=50) assigned to standard care (all subjects will be offered a 3-month supply of nicotine replacement therapy) and (4) to conduct exploratory analyses of putative moderators and mediators of program efficacy.

If the mobile version of PSF is proven to be feasible and efficacious, the project will have short term impact by opening a new vista of tobacco (and other behavioral) treatment for a highly vulnerable group. Study data will provide crucial information for a definitive trial of the intervention. The long-term impact will be reduced tobacco-related morbidity and mortality among PLWH, and a clearer understanding of the role of mHealth in comprehensive HIV care.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Current cigarette smoker
* Has a smartphone
* Interested in quitting
* Receives care at the Montefiore Center for Positive Living

Exclusion Criteria:

* Pregnancy
* Contraindication to nicotine patch use
* Fails to meet inclusion criteria above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Biochemically-verified (by exhaled breath carbon-monoxide level), 7-day point-prevalence-abstinence at the 3 month timepoint | 3-months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Background] Shuter J, Morales DA, Considine-Dunn SE, An LC, Stanton CA. Feasibility and preliminary efficacy of a web-based smoking cessation intervention for HIV-infected smokers: a randomized controlled trial. J Acquir Immune Defic Syndr. 2014 Sep 1;67(1):59-66. doi: 10.1097/QAI.0000000000000226. PMID 25118794